CLINICAL TRIAL: NCT05133076
Title: A Randomized Placebo-controlled Study to Assess Safety and Preliminary Efficacy of BGP345A in Patients With Constipation Due to the Use of Opioid-based Medications for the Management of Chronic Non Cancer Pain
Brief Title: Safety and Preliminary Efficacy of BGP345A in Constipation Due to Opioid-based Medications
Acronym: OIC1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioGaia Pharma AB (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEC19156
Record Dates: First submitted 2021-10-26; First posted 2021-11-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2023-09

CONDITIONS: Opioid-Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm (Active Comparator)
  Interventions: Biological: Lactobacillus gasseri BGP345A
- Placebo arm (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus gasseri BGP345A — Active and placebo capsules for oral use
  Other Names: BGP345A
  Arms: Active arm
Biological: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to assess safety and preliminary efficacy of BGP345A in patients with constipation due to the use of opioid-based medications for the management of chronic non cancer pain.

ELIGIBILITY:
Inclusion Criteria:

I1. Age over 18 years (limit included),

I2. Diagnosed with OIC according to the adapted ROME IV criteria (Mearin F et al, 2016) previously used in clinical evaluation of patients with OIC (Webster LR et al, 2017) and self-reported symptoms assessed by a physician (daily diary check at V1 visit):

* Fewer than three (<3) spontaneous bowel movements (SBMs) per week. A SBM is defined as a bowel movement without the use of laxatives in the previous 24 hours as recorded in the daily diary.
* And one or more of the following symptoms in at least 25% of bowel movements: straining, feeling of incomplete evacuation, and/or hard/small stools, defined as Bristol Stool Scale (BSS) score lower than 3 (<3).

I3. With chronic non-cancer pain since at least three months, including the following indications but not limited to: back-pain, rheumatisms and post-operative pain,

I4. Patients received opioids for chronic analgesia (intended treatment ≥6 Weeks) for 1 week or more prior to study start and a stable regimen of opioids for 3 or more days before study entry (V0 visit) and during the whole study ,

I5. Subjects must be willing to discontinue laxative use at screening and only use the rescue laxatives permitted throughout the study duration,

I6. For women:

* Non menopausal with the same reliable contraception since at least 2 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study (condom with spermicide gel, any oral contraceptive, intrauterine device, subcutaneous contraceptive implant, vaginal ring, surgical intervention (bilateral tubal ligation or ovariectomy or hysterectomy), ESSURE system),
* Menopausal without or with hormone replacement therapy,

I7. Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,

I8. Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,

I9. Affiliated with a social security scheme.

Exclusion Criteria:

E1. Involvement in any investigational drug or device study within 30 days prior to this study,

E2. Unable to withdraw other OIC treatments (any kind of laxative other than provided in the study),

E3. History of chronic constipation prior to starting analgesic medication or any potential non-opioid cause of bowel dysfunction that may be a major contributor to the constipation upon investigator judgment,

E4. Surgery planned within the whole study period,

E5. Evidence of active medical diseases affecting bowel transit,

E6. Antibiotic treatment intake within the last month prior the study start (V0),

E7. Unwilling to withdraw probiotic supplements, yoghurts without supplemented bacteria are permitted,

E8. Any history of drug addiction in the past five years,

E9. Pregnant or lactating women or intending to become pregnant,

E10. Unwilling to maintain food habits and current physical activity for the whole study duration,

E11. With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,

E12. Having a lifestyle deemed incompatible with the study according to the investigator including drug and alcohol abuse,

E13. Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,

E14. Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,

E15. Presenting a psychological or linguistic incapability to sign the informed consent,

E16. Impossible to contact in case of emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Change in the average weekly number of Spontaneous Bowel Movements (SBMs) (expressed in number of stools/week) | Over the 4 week treatment period
  A SBM (Spontaneous Bowel Movement) is defined as a bowel movement without the use of laxatives in the previous 24 hours as recorded in the daily diary (Webster LR et al, 2017).

SECONDARY OUTCOMES:
Percentage of responders over the 4-weeks of treatment period defined by subjects reporting an average weekly number of SBMs ≥ 3 and an increase of the average weekly number of SBM ≥1 from baseline | Average over the last two weeks of treatment
  SBM responders
Change in the average weekly number of BMs (Bowel Movements) | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  BM (Bowel Movements) expressed in number of stools/week
Change in the average weekly number of CSBMs (Complete Spontaneous Bowel Movement) | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  CSBMs (Complete Spontaneous Bowel Movement) expressed in number of stools/week is defined by as a bowel movement without the use of laxatives in the previous 24 hours as recorded in the daily diary and the feeling of complete emptying after bowel movement.
Change in the average weekly number of SBMs | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  SBMs expressed in number of stools/week
Change in the average weekly number of SBMs with no straining (straining score 1) | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  SBMs expressed in number of stools/week
Time to first SBM and CSBM after the last recorded stool before the randomisation | Over 4 week treatment period
  Expressed in hours
Change in the number of days with presence of SBMs | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  SBMs expressed in days/week
Change in the number of days with presence of CSBMs | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  CSBMs expressed in days/week
Change in the average weekly number of SBMs rated 3 or 4 on the BSS (Bristol Stool Scale) | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  Expressed in stools/week
Change of stool consistency assessed by the BSS (Bristol Stool Scale) | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  Expressed in arbitrary units/stool from 1-7.
Change of the overall BFI (Bowel Function Index) score | Over 4 week treatment period
  Expressed in arbitrary units, range 0-100
Change in the average daily abdominal bloating score | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  Expressed in arbitrary units/day (this score will be assessed daily for the past 24hours and could range from 0 to 4, where 0 = absent or no bloating, 1 = mild, 2 = moderate, 3= severe, and 4 =very severe bloating)
Change in the average daily abdominal discomfort score | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  Expressed in arbitrary units/day (this score will be assessed daily for the past 24hours and could range from 0 to 4, where 0 = no abdominal discomfort, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe discomfort)
Change in average daily pain at defecation assessed by the Visual Analogic Scale for pain at defecation (VAS) | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  Expressed in arbitrary units/day with stool, range 0-100
Change in the weekly frequency of rescue laxative use assessed by the daily diary | Over 4 week treatment period; during each week of the treatment period; and up to 8 weeks at study completion.
  expressed in average of days/week
Frequency of rescue laxative use assessed by the daily diary. | Over the 4 week treatment period
  Expressed in number of laxative uses
General health state measuring vital parameters assessed - Body weight | Through study completion, 10 weeks
  Body weight (kg)
General health state measuring vital parameters assessed- Diastolic Blood Pressure | Through study completion, 10 weeks
  Diastolic Blood Pressure (mmHg)
General health state measuring vital parameters assessed- Systolic Blood Pressure | Through study completion, 10 weeks
  Systolic Blood Pressure (mmHg)
General health state measuring vital parameters assessed- Vital signs | Through study completion, 10 weeks
  Vital signs (BPM)
the frequency of adverse events (AE), serious adverse events (SAE), Treatment-Emergent Adverse events (TEAE), Serious treatment-emergent adverse events (STEAE) | Through study completion, 10 weeks
  Frequency and nature of events

CONTACTS AND LOCATIONS:
Overall Officials: Petra J Lierud, Study Director — BioGaia Pharma
Locations (4):
- France (4):
  - Groupe hospitalier Saint-Joseph, Paris, Paris
  - CHU d'Amiens, Amiens
  - CHU DE NANTES (Hôpital Nord Laennec), Saint-Herblain
  - CH de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No